CLINICAL TRIAL: NCT05572515
Title: A Phase 3 Randomized Study Comparing Teclistamab Monotherapy Versus Pomalidomide, Bortezomib, Dexamethasone (PVd) or Carfilzomib, Dexamethasone (Kd) in Participants With Relapsed or Refractory Multiple Myeloma Who Have Received 1 to 3 Prior Lines of Therapy, Including an Anti-CD38 Monoclonal Antibody and Lenalidomide
Brief Title: A Study Comparing Teclistamab Monotherapy Versus Pomalidomide, Bortezomib, Dexamethasone (PVd) or Carfilzomib, Dexamethasone (Kd) in Participants With Relapsed or Refractory Multiple Myeloma
Acronym: MajesTEC-9
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR109244; 64007957MMY3006 (Other: Janssen Research & Development, LLC); 2022-000928-37 (EudraCT Number); 2023-503444-13-00 (Registry Identifier: EUCT number)
Expanded Access: NCT05463939 (Approved for marketing)
Record Dates: First submitted 2022-10-05; First posted 2022-10-07 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Relapsed or Refractory Multiple Myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma | interventions — pomalidomide; Bortezomib; Dexamethasone; carfilzomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Teclistamab (Experimental): Participants will receive teclistamab monotherapy in Part 1 and an alternative dosing regimen of teclistamab in Part 2.
  Interventions: Drug: Teclistamab
- Pomalidomide, Bortezomib and Dexamethasone (PVd) or Carfilzomib and Dexamethasone (Kd) (Experimental): Participants will receive either PVd or Kd based on principal investigator's choice during Part 1 of the study.
  Interventions: Drug: Pomalidomide; Drug: Bortezomib; Drug: Dexamethasone; Drug: Carfilzomib

INTERVENTIONS:
Drug: Teclistamab — Teclistamab will be administered subcutaneously.
  Other Names: JNJ-64007957
  Arms: Teclistamab
Drug: Pomalidomide — Pomalidomide will be administered orally.
  Arms: Pomalidomide, Bortezomib and Dexamethasone (PVd) or Carfilzomib and Dexamethasone (Kd)
Drug: Bortezomib — Bortezomib will be administered subcutaneously.
  Arms: Pomalidomide, Bortezomib and Dexamethasone (PVd) or Carfilzomib and Dexamethasone (Kd)
Drug: Dexamethasone — Dexamethasone will be administered orally in PVd and intravenously or orally in Kd.
  Arms: Pomalidomide, Bortezomib and Dexamethasone (PVd) or Carfilzomib and Dexamethasone (Kd)
Drug: Carfilzomib — Carfilzomib will be administered intravenously.
  Arms: Pomalidomide, Bortezomib and Dexamethasone (PVd) or Carfilzomib and Dexamethasone (Kd)

SUMMARY:
The purpose of this study is to compare the efficacy of teclistamab with PVd/Kd in Part 1 and to further characterize safety and efficacy of an alternative dosing for teclistamab in Part 2 in participants with relapsed or refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of multiple myeloma as defined by the criteria below: (a)Multiple myeloma diagnosis according to International Myeloma Working Group (IMWG) diagnostic criteria (b) Measurable disease at screening as defined by any of the following: (1) Serum M-protein level greater than or equal to (>=)0.5 grams per deciliter (g/dL) (central laboratory); or (2) Urine M-protein level >=200 milligrams (mg)/24 hours (central laboratory); or (3) Serum immunoglobulin free light chain >=10 milligrams per deciliter (mg/dL) (central laboratory) and abnormal serum immunoglobulin kappa lambda free light chain ratio
* Received 1 to 3 prior lines of antimyeloma therapy including a minimum of 2 consecutive cycles of an anti- cluster of differentiation 38 (CD38) monoclonal antibody at the approved dosing regimen in any prior line and 2 consecutive cycles of lenalidomide in any prior line
* Documented evidence of progressive disease or failure to achieve a response to last line of therapy based on investigator's determination of response by International myeloma working group (IMWG) criteria
* Have an Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 2
* A female participant must agree not to be pregnant, breast-feeding, or plan to become pregnant while enrolled in this study or within 6 months after the last dose of study treatment
* Must be willing and able to adhere to the lifestyle restrictions specified in this protocol

Exclusion Criteria:

* Received any prior B cell maturation antigen (BCMA)-directed therapy
* A participant is not eligible to receive PVd as control therapy if any of the following are present: (1) Received prior pomalidomide therapy, (2) Does not meet criteria for bortezomib retreatment (3) Contraindications or life-threatening allergies, hypersensitivity, or intolerance to pomalidomide or bortezomib, (4) Grade 1 peripheral neuropathy with pain or Grade greater than or equal to (>=) 2 peripheral neuropathy as defined by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0, (5) Received a strong cytochrome P (CYP) 3A4 inducer within 5 half-lives prior to randomization; A participant is not eligible to receive Kd as control therapy if any of the following are present:(1) Received prior carfilzomib therapy, (2) Uncontrolled hypertension, defined as an average systolic blood pressure greater than (>)159 millimeters of mercury (mmHg) or diastolic blood pressure >99 mmHg despite optimal treatment (3) Grade 2 peripheral neuropathy with pain or Grade >=3 peripheral neuropathy as defined by NCI-CTCAE Version 5.0, (4) Contraindications or life-threatening allergies, hypersensitivity, or intolerance to carfilzomib (intolerance defined as prior therapy discontinued due to any adverse event [AE] related to carfilzomib)
* Received a maximum cumulative dose of corticosteroids of >=140 mg of prednisone or equivalent within 14 days prior to randomization
* Received a live, attenuated vaccine within 4 weeks before randomization
* Central nervous system (CNS) involvement or clinical signs of meningeal involvement of multiple myeloma
* Plasma cell leukemia at the time of screening, Waldenstrom's macroglobulinemia, polyneuropathy, organomegaly, endocrinopathy, M-protein (POEMS) syndrome and skin changes, or primary amyloid light chain amyloidosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 614 (Actual)
Dates: Start 2023-03-29 (Actual); Primary Completion 2026-02-13 (Estimated); Study Completion 2031-08-31 (Estimated)

PRIMARY OUTCOMES:
Part 1: Progression-free Survival (PFS) | Up to 9 years
  PFS is defined as the time from the date of randomization to the date of first documented disease progression, as defined in the International myeloma working group (IMWG) 2016 response criteria, or death due to any cause, whichever occurs first.
Part 2: Number of Participants Reporting Cytokine Release Syndrome (CRS) Cases by Severity | Up to 9 years
  Severity for CRS will be graded as follows: Grade 1: Fever (Temperature greater than or equal to [>=] 38°C); Grade 2: Fever (Temperature >=38°C) with either: hypotension and/or hypoxia requiring low-flow nasal cannula or blow-by; Grade 3: Fever (Temperature >=38°C) with either: hypotension and/or hypoxia requiring high-flow nasal cannula, facemask, nonrebreather mask, or Venturi mask; Grade 4: Fever (Temperature >=38°C) with either: hypotension requiring multiple vasopressors (excluding vasopressin), and/or hypoxia requiring positive pressure and Grade 5: Death.

SECONDARY OUTCOMES:
Part 1 and 2: Overall Response (Partial Response [PR] or Better) | Up to 9 years
  Overall response (PR or better) is defined as participants who have a PR or better prior to subsequent antimyeloma therapy in accordance with the IMWG 2016 criteria.
Part 1 and 2: Very Good Partial Response (VGPR) or Better Response | Up to 9 years
  VGPR or better (Stringent Complete Response [sCR]+Complete Response [CR]+VGPR) is defined as participants who achieve a VGPR or better response prior to subsequent antimyeloma therapy in accordance with the IMWG 2016 criteria.
Part 1 and 2: Complete Response (CR) or Better Response | Up to 9 years
  CR or better response is defined as participants who achieve a CR or better response prior to subsequent antimyeloma therapy in accordance with the IMWG 2016 criteria.
Part 1: Duration of Response (DOR) | Up to 9 years
  DOR is defined as the time interval between the date of initial documentation of a response (PR or better) to the date of first documented evidence of progressive disease according to the IMWG 2016 response criteria or death due to any cause, whichever occurs first.
Part 1: Time to Next Treatment (TTNT) | Up to 9 years
  TTNT is defined as the time from randomization to the start of subsequent antimyeloma treatment.
Part 1: Progression-free Survival on Next-line Therapy (PFS2) | Up to 9 years
  PFS2 is defined as the time interval between the date of randomization and date of event, which is defined as progressive disease as assessed by investigator on the first subsequent line of antimyeloma therapy, or death from any cause, whichever occurs first.
Part 1: Overall Survival (OS) | Up to 9 years
  OS is defined as the time from the date of randomization to the date of the participant's death due to any cause.
Part 1 and 2: Number of Participants with Adverse Events (AEs) by Severity | Up to 9 years
  Number of participants with AEs by Severity will be reported.
Part 1 and 2: Number of Participants with Serious Adverse Events (SAEs) by Severity | Up to 9 years
  Number of participants with SAEs by Severity will be reported.
Part 1 and 2: Number of Participants with Abnormal Laboratory Results | Up to 9 years
  Number of participants with abnormal laboratory results (such as hematology and chemistry) will be reported.
Part 1 and 2: Serum Concentrations of Teclistamab | Up to 9 years
  Serum concentrations of teclistamab will be reported.
Part 1 and 2: Number of Participants with Anti-drug Antibodies (ADAs) to Teclistamab | Up to 9 years
  Number of participants with ADAs to teclistamab will be reported.
Part 1: Change from Baseline in Symptoms, Functioning, and Overall Health-related Quality of Life (HRQoL) as Assessed by European Organization for Research and Treatment of Cancer Quality-of-life Questionnaire Core 30 (EORTC-QLQ-C30) | Baseline up to 9 years
  Change from baseline in symptoms, functioning, and overall HRQoL assessed by EORTC QLQ-C30 score version 3 will be reported. The EORTC- QLQ-C30 Version 3 includes 30 items that make up 5 functional scales (physical, role, emotional, cognitive, and social), 1 global health status scale, 3 symptom scales (pain, fatigue, and nausea/vomiting), and 6 single symptom items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The item and scale scores are transformed to a 0 to 100 scale. A high scale score represents a higher response level. Thus, a high score for a functional scale represents a high/healthy level of functioning and a high score for the global health status represents high HRQoL, but a high score for a symptom scale/item represents a high level of symptomatology/problems.
Part 1: Change from Baseline in Symptoms, Functioning, and Overall HRQoL as Assessed by Multiple Myeloma Symptom and Impact Questionnaire (MySIm-Q) Scale Score | Baseline up to 9 years
  Change from baseline in symptoms, functioning, and overall HRQoL assessed by MySIm-Q will be reported. The MySIm-Q is a disease-specific PRO assessment complementary to the EORTC-QLQ-C30. It includes 17 items resulting in a symptom subscale and an impact subscale. The recall period is the "past 7 days", and responses are reported on a 5-point verbal rating scale.
Part 1: Change from Baseline in Symptoms, Functioning, and Overall HRQoL as Assessed by Patient-reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) | Baseline up to 9 years
  Change from baseline in symptoms, functioning, and overall HRQoL assessed by PRO-CTCAE will be reported. The National Cancer Institute's (NCI's) PRO-CTCAE is an item library of common adverse events experienced by people with cancer that are appropriate for self-reporting of treatment tolerability. Each symptom selected for inclusion can be rated by up to 3 attributes characterizing the presence/frequency, severity, and/or interference of the AEs. It ranges from 0 to 4 with higher scores indicating higher frequency or greater severity/impact.
Part 1: Change from Baseline in Symptoms, Functioning, and Overall HRQoL as Assessed by EuroQol Five Dimension Questionnaire 5-Level (EQ-5D-5L) | Baseline up to 9 years
  Change from baseline in symptoms, functioning, and overall HRQoL assessed by EQ-5D-5L will be reported. The EQ-5D-5L is a generic measure of health status. The EQ-5D-5L is a 5-item questionnaire that assesses 5 domains including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression plus a visual analog scale rating "health today" with anchors ranging from 0 (worst imaginable health state) to 100 (best imaginable health state).
Part 1: Time to Worsening in Symptoms, Functioning, and Overall HRQoL | Up to 9 years
  Time to worsening in symptoms, functioning, and overall HRQoL will be measured as the interval from the date of randomization to the start date of meaningful change.
Part 1: PFS in Participants in High-risk Molecular Features | Up to 9 years
  PFS in participants in high-risk molecular features will be reported. PFS is defined as the time from the date of randomization to the date of first documented disease progression, as defined in the IMWG 2016 response criteria, or death due to any cause, whichever occurs first.
Part 1: Depth of Response in Participants in High-risk Molecular Features | Up to 9 years
  Depth of response in participants in high-risk molecular features will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (210):
- United States (30):
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Alta Bates Comprehensive Cancer Center, Berkeley, California
  - MemorialCare Long Beach Medical Center, Long Beach, California
  - University of California Irvine, Orange, California
  - PIH Health Hospital, Whittier, California
  - Rocky Mountain Cancer Centers, Aurora, Colorado
  - University of Connecticut, Farmington, Connecticut
  - University of Miami Sylvester Cancer Center, Miami, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Mission Cancer Blood, Waukee, Iowa
  - East Jefferson General Hospital Bone Marrow Transport Clinic, Metairie, Louisiana
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Maryland Oncology Hematology P A, Silver Spring, Maryland
  - Boston University Medical Center, Boston, Massachusetts
  - Saint Lukes Hospital Saint Lukes Cancer Specialists, Chesterfield, Missouri
  - Cooper Health System MD Anderson Cancer Center at Cooper, Camden, New Jersey
  - Herbert Irving Comprehensive Cancer Center Columbia University Medical Center, New York, New York
  - Durham VAMC, Durham, North Carolina
  - Penn Medicine Lancaster General Health, Lancaster, Pennsylvania
  - Tennessee Oncology, Nashville, Tennessee
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Michael E DeBakey VA Medical Center, Houston, Texas
  - Harris Health Smith Clinic, Houston, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Alexander T. Augusta Military Medical Center, Fort Belvoir, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - NorthWest Medical Specialties, PLLC, Tacoma, Washington
- Australia (5):
  - Blacktown Hospital, Blacktown
  - St Vincents Hospital Melbourne, Fitzroy
  - Box Hill Hospital, Melbourne
  - Fiona Stanley Hospital, Murdoch
  - Sir Charles Gairdner Hospital, Nedlands
- Austria (2):
  - LKH - Universitätsklinikum der PMU Salzburg, Salzburg
  - Medical University Vienna MUV, Vienna
- Belgium (5):
  - Algemeen Ziekenhuis Klina, Brasschaat
  - Jolimont, Haine-St-Paul
  - Az Groeninge, Kortrijk
  - Universitair Ziekenhuis Gasthuisberg, Leuven
  - CHR de la Citadelle, Liège
- Brazil (16):
  - Hospitais Integradaos da Gavea S/A - DF Star, Brasília
  - Fundacao Universidade de Caxias do Sul, Caxias do Sul
  - Liga Paranaense de Combate ao Cancer, Curitiba
  - Instituto Joinvilense de Hematologia e Oncologia Ltda Centro de Hematologia e Oncologia, Joinville
  - Liga Norte Riograndense Contra O Cancer, Natal
  - Complexo Hospitalar de Niteroi, Niterói
  - Instituto de Educacao, Pesquisa e Gestao em Saude Instituto Americas (COI), Rio de Janeiro
  - Hospital Sao Rafael, Salvador
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto Hospital de Base, São José do Rio Preto
  - Sociedade Beneficente de Senhoras Hospital Sirio Libanes, São Paulo
  - Real e Benemérita Associação Portuguesa de Beneficência, São Paulo
  - Hospital Alemao Oswaldo Cruz, São Paulo
  - Instituto D Or de Pesquisa e Ensino IDOR, São Paulo
  - Fundacao Antonio Prudente A C Camargo Cancer Center, São Paulo
  - Clinica Medica Sao Germano LTDA, São Paulo
  - Sociedade Beneficente Israelita Brasileira Hospital Albert Einstein, São Paulo
- Canada (5):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Brampton Civic Hospital, Brampton, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - CIUSSS de l Est de l Ile de Montreal Installation Hopital Maisonneuve Rosemont, Montreal, Quebec
- China (23):
  - Beijing Chaoyang Hospital, Beijing
  - BeiJing JiShuiTan Hospital, Beijing
  - The First Bethune Hospital of Jilin University, Changchun
  - The Third Xiangya Hospital, Central South University, Changsha
  - Sichuan Provincial Peoples Hospital, Chengdu
  - Chongqing University Cancer Hospital, Chongqing
  - Fujian Meidical University Union Hospital, Fuzhou
  - Sun Yat -Sen University Cancer Center, Guangzhou
  - First affiliated Hospital of Zhejiang University, Hangzhou
  - Harbin medical university cancer hospital, Harbin
  - The First Affiliated Hospital of NanChang University, Nanchang
  - Nanjing Drum Tower Hospital, Nanjing
  - First Affiliated Hospital of Guangxi Medical University, Nanning
  - Shanghai Fourth People s Hospital, Shanghai
  - Shengjing Hospital Of China Medical University, Shenyang
  - Shenzhen 2nd People's Hospital, Shenzhen
  - Institute of Hematology and Blood Diseases Hospital, Tianjin
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - Wuhan Union Hospital, Wuhan
  - Wuxi People s Hospital, Wuxi
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - Henan Cancer Hospital, Zhengzhou
- Czechia (4):
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni Nemocnice Ostrava, Ostrava - Poruba
  - Vseobecna fakultni nemocnice v Praze, Prague
- Denmark (6):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Regionshospitalet Godstrup, Herning
  - Odense Universitetshospital, Odense C
  - Vejle Sygehus, Vejle
- France (12):
  - CHU Amiens - Hopital Sud, Amiens
  - Hôpital Côte de Nacre, Caen
  - CHU Grenoble, Grenoble
  - Centre Hospitalier du Mans, Le Mans
  - Hopital Saint Vincent de Paul, Lille
  - CHU de Montpellier Hopital Saint Eloi, Montpellier
  - CHU Nantes, Nantes
  - Hopital Saint-Antoine, Paris
  - Hopital de la Pitie Salpetriere, Paris
  - Hopital Necker Enfants Malades, Paris
  - Institut Universitaire du Cancer Toulouse Oncopole, Toulouse
  - CHU de Nancy - Hopital de Brabois, Vandœuvre-lès-Nancy
- Germany (9):
  - Medizinische Universitat Lausitz Carl Thiem, Cottbus
  - Universitatsklinikum Carl Gustav Carus Dresden, Dresden
  - Universitätsmedizin Greifswald, Greifswald
  - Asklepios Klinik Altona, Hamburg
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum Giessen und Marburg GmbH, Marburg
  - Universitatsklinikum Tubingen, Tübingen
  - Universitatsklinikum Ulm, Ulm
  - Heinrich-Braun-Klinikum gGmbH, Zwickau
- Greece (3):
  - Alexandra General Hospital of Athens, Athens Attica
  - Agios Andreas General Hospital of Patra, Pátrai
  - G Papanikolaou Hospital of Thessaloniki, Thessaloniki
- India (3):
  - Fortis Memorial Research Institute, Gūrgaon
  - Bhagwan Mahaveer Cancer Hospital & Research Centre, Jaipur
  - Deenanath Mangeshkar Hospital and Research Centre, Pune
- Israel (6):
  - Hillel Yaffe Medical Center, Hadera
  - Bnai Zion Medical Center, Haifa
  - Carmel Medical Center, Haifa
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (10):
  - A O U Sant Orsola Malpighi, Bologna
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Azienda Ospedaliero Universitaria Policlinico Paolo Giaccone, Palermo
  - Ospedale Santa Chiara AO Universitaria Pisana, Pisa
  - Arcispedale Santa Maria Nuova - IRCCS, Reggio Emilia
  - Campus Bio Medico di Roma, Roma
  - A O Universitaria Senese Ospedale Santa Maria alle Scotte, Siena
  - A.O.U. Citta della Salute e della Scienza di Torino - Presidio Molinette, Turin
  - ASUI Santa Maria della Misericordia di Udine, Udine
  - Ospedale di Circolo e Fondazione Macchi, Varese
- Japan (21):
  - Institute of Science Tokyo Hospital, Bunkyō City
  - Chiba Cancer Center, Chiba
  - Ogaki Municipal Hospital, Gifu
  - National Hospital Organization Shibukawa Medical Center, Gunma
  - Kansai Medical University Hospital, Hirakata
  - Hitachi General Hospital, Hitachi
  - Saitama Medical University Hospital, Iruma-gun
  - Kameda Medical Center, Kamogawa
  - National Cancer Center Hospital East, Kashiwa
  - Kurashiki Central Hospital, Kurashiki
  - Matsuyama Red Cross Hospital, Matsuyama
  - Aichi Medical University Hospital, Nagakute
  - JRC Nagasaki Genbaku Hospital, Nagasaki
  - Niigata University Medical And Dental Hospital, Niigata
  - National Hospital Organization Okayama Medical Center, Okayama
  - Osaka Metropolitan University Hospital, Osaka
  - Hokkaido University Hospital, Sapporo
  - Juntendo University Hospital, Tokyo
  - The Cancer Institute Hospital of JFCR, Tokyo
  - Yamagata University Hospital, Yamagata
  - Yamanashi Prefectural Central Hospital, Yamanashi
- Malaysia (4):
  - Hospital Pulau Pinang, George Town
  - Hospital Queen Elizabeth, Kota Kinabalu
  - University Malaya Medical Centre, Kuala Lumpur
  - Subang Jaya Medical Centre, Subang Jaya
- Netherlands (4):
  - Meander Medisch Centrum, Amersfoort
  - VUMC Amsterdam, Amsterdam
  - Universitair Medisch Centrum Groningen, Groningen
  - UMC Utrecht, Utrecht
- Poland (4):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Pratia Onkologia Katowice, Katowice
  - Swietokrzyskie Centrum Onkologii SPZOZ w Kielcach, Kielce
  - Uniwersytecki Szpital Kliniczny Nr 1 w Lublinie, Lublin
- Portugal (5):
  - Uls Almada Seixal - Hosp. Garcia de Orta, Almada
  - Uls Braga - Hosp. Braga, Braga
  - Champalimaud Foundation Champalimaud Centre, Lisbon
  - Instituto Portugues de Oncologia, Porto
  - Uls Gaia Espinho, Vila Nova de Gaia
- Spain (13):
  - Hosp. Univ. Germans Trias I Pujol, Badalona
  - Hosp. de Jerez de La Frontera, Jerez de la Frontera
  - Institut Catala d Oncologia L Hospitalet, L'Hospitalet de Llobregat
  - Hosp. de Leon, León
  - Hosp. Univ. Infanta Leonor, Madrid
  - Hosp. Univ. Ramon Y Cajal, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Gral. Univ. J.M. Morales Meseguer, Murcia
  - Hospital Universitario Central de Asturias, Oviedo
  - Hosp. Son Llatzer, Palma de Mallorca
  - Hosp. Montecelo, Pontevedra
  - Hosp. Quiron Madrid Pozuelo, Pozuelo de Alarcón
  - Hospital Universitari i Politecnic La Fe, Valencia
- Sweden (3):
  - Falu Lasarett Medicinkliniken Falun, Falun
  - Helsingborgs lasarett, Helsingborg
  - Akademiska Sjukhuset, Uppsala
- Turkey (Türkiye) (8):
  - Ankara Gulhane Training and Research Hospital, Ankara
  - Dr Abdurrahman Yurtaslan Oncology Training and Research Hospital, Ankara
  - Ankara University Medical Faculty, Ankara
  - Liv Hospital Ankara, Ankara
  - Antalya Training And Research Hospital, Antalya
  - Ondokuz Mayis University, Atakum
  - Pamukkale University Medical Faculty, Denizli
  - Medipol University Hospital, Istanbul
- United Kingdom (9):
  - Aberdeen Royal Infirmary, Aberdeen
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Colchester Hospital University NHS, Colchester
  - The Clatterbridge Cancer Centre, Liverpool
  - Chelsea And Westminster Hospital, London
  - St Georges Hospital, London
  - James Cook University Hospital, Middlesbrough
  - Norfolk and Norwich University Hospital, Norwich
  - Royal Stoke University Hospital, Staffordshire

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency